CLINICAL TRIAL: NCT04496492
Title: Preoperative Use of Tocotrienol Associated With Personalized Nutritional and Psychoeducational Support in Women With Primary Breast Cancer.
Brief Title: Preoperative Use of Tocotrienol From Annatto Bixa Orellana L. in Breast Cancer Patients: a Prospective Clinical Trial.
Acronym: TOCANNATO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-005275-92
Record Dates: First submitted 2020-06-26; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tocotrienols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocotrienol (Experimental): Subjects receiveTocotrienol 200 mg/twice daily before surgery
  Interventions: Drug: Tocotrienol

INTERVENTIONS:
Drug: Tocotrienol — Tocotrienol 200 mg orally twice a day

SUMMARY:
Tocotrienols have shown strong in vitro and in vivo anti-oxidant and anticancer activity, promoting apoptosis and regulating oncogenic targets in breast cancer. However their clinical use is still experimental especially in preoperative setting, where there are still no data of antioxidant and antiinflammatory beneficial roles. This study is a prospective observational clinical study enrolling 50 patients with primary breast cancer (T1-2, N0-1, M0) who received 4-weeks oral treatment of delta-T3 before surgery (200 mg/twice daily) with personalized nutritional and psychoeducational support. This study evaluates the effects of treatment on oxidant (tock fast-Li Starfish) and antioxidant capacity (TAC Track, Li Starfish), anti-inflammatory activity (complete profiling of adaptive and innate cell immunity, immunologic serum markers (miRNA)), immunological response on tumor (gene expression profiling on preoperative tissue tumor biopsy and on surgical specimen), TNF-alpha, IL-6 and VEGF and proliferation/apoptosis, anti-inflammatory and anti-oxidant activity of breast cancer cell lines.

This study evaluates the effects of treatment on oxidant (tock fast-Li Starfish) and antioxidant capacity (TAC Track, Li Starfish), on anti-inflammatory activity (complete profiling of adaptive and innate cell immunity, immunologic serum markers (miRNA)), on immunological response on tumor (gene expression profiling on preoperative tissue tumor biopsy and on surgical specimen), on TNF-alpha, IL-6 and VEGF, on proliferation/apoptosis, anti-inflammatory and anti-oxidant activity of breast cancer cell lines.

DETAILED DESCRIPTION:
An open-label, single center, phase 2 prospective observational clinical study

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed operable primary breast cancer (T1-T2 N0-1 M0)
* absence of distant metastasis
* signed informed consent.

Exclusion Criteria:

* Previous malignancies other than in situ cervical carcinoma or nonmelanoma skin cancer
* Breast cancer recurrence
* Metastatic breast cancer
* Non-epithelial breast cancer at histological examination
* In situ lobular breast cancer
* Participation in other randomized clinical trials that could interfere with current study
* Living distant from center and unable to attend for check-ups and meetings

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Changes in blood oxidant capacity | 4 weeks
  Oxidant capacity (through tock fast-Li Starfish) (µmol/L) was measured in patients' serum samples.
Changes in blood antioxidant capacity | 4 weeks
  Antioxidant capacity (through TAC Track, Li Starfish) (µmol/L) was measured in patients' serum samples.
Absolute and relative changes in peripheral blood mononuclear cells obtained before and after four weeks of tocotrienol treatment, as detected by 13-colors citofluorimetry analysis | 4 weeks
  Peripheral blood mononuclear cells were measured by 13-color cytofluorimetry analysis in patients' serum samples.
Changes of immune-related miRNA levels in patients' serum samples obtained before and after four weeks of tocotrienol treatment, as determined by quantitative real-time PCR analysis | 4 weeks
  Immune-related miRNA levels were determined by quantitative real-time PCR analysis in patients' serum samples obtained before and after four weeks of tocotrienol treatment
Changes in immune response associated gene levels in preoperative tissue tumor biopsies and in surgical specimens, obtained before and after four weeks of tocotrienol treatment, respectively, as determined by gene expression profiling analysis | 4 weeks
  Immune response associated gene levels were determined by gene expression profiling analysis in preoperative tissue tumor biopsies and in surgical specimens, obtained before and after four weeks of tocotrienol treatment
Changes in serum inflammatory cytokines and growth factor | 4 weeks
  Blood inflammatory cytokines and growth factor (through TNF-alpha (pg/ml), IL-6 (pg/ml) and VEGF (pg/ml) quantifications) were measured in patients' serum samples

SECONDARY OUTCOMES:
Treatment-induced changes in proliferation/apoptosis, anti-inflammatory and anti-oxidant activity of breast cancer cell lines | 12,24 and 72 hours
  Treatment-induced changes in proliferation/apoptosis, anti-inflammatory and anti-oxidant activity of breast cancer cell lines was measured through cell culture analysis.
Changes in expression of tumor proliferation, hormone receptors and HER2 | 4 weeks
  Expression of tumor proliferation index (Ki67), estrogen and/progesterone receptor and HER2 oncoprotein by IHC was determined in preoperative tumor biopsies and in surgical specimens

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ferraris, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

REFERENCES:
- [Result] Qureshi AA, Pearce BC, Nor RM, Gapor A, Peterson DM, Elson CE. Dietary alpha-tocopherol attenuates the impact of gamma-tocotrienol on hepatic 3-hydroxy-3-methylglutaryl coenzyme A reductase activity in chickens. J Nutr. 1996 Feb;126(2):389-94. doi: 10.1093/jn/126.2.389. PMID 8632210
- [Result] Rasool AH, Rahman AR, Yuen KH, Wong AR. Arterial compliance and vitamin E blood levels with a self emulsifying preparation of tocotrienol rich vitamin E. Arch Pharm Res. 2008 Sep;31(9):1212-7. doi: 10.1007/s12272-001-1291-5. Epub 2008 Sep 20. PMID 18806966
- [Result] Song BL, DeBose-Boyd RA. Insig-dependent ubiquitination and degradation of 3-hydroxy-3-methylglutaryl coenzyme a reductase stimulated by delta- and gamma-tocotrienols. J Biol Chem. 2006 Sep 1;281(35):25054-61. doi: 10.1074/jbc.M605575200. Epub 2006 Jul 10. PMID 16831864
- [Result] Pearce BC, Parker RA, Deason ME, Qureshi AA, Wright JJ. Hypocholesterolemic activity of synthetic and natural tocotrienols. J Med Chem. 1992 Oct 2;35(20):3595-606. doi: 10.1021/jm00098a002. PMID 1433170
- [Result] Begum AN, Terao J. Protective effect of alpha-tocotrienol against free radical-induced impairment of erythrocyte deformability. Biosci Biotechnol Biochem. 2002 Feb;66(2):398-403. doi: 10.1271/bbb.66.398. PMID 11999415
- [Result] Palozza P, Verdecchia S, Avanzi L, Vertuani S, Serini S, Iannone A, Manfredini S. Comparative antioxidant activity of tocotrienols and the novel chromanyl-polyisoprenyl molecule FeAox-6 in isolated membranes and intact cells. Mol Cell Biochem. 2006 Jul;287(1-2):21-32. doi: 10.1007/s11010-005-9020-7. Epub 2006 Apr 28. PMID 16645729
- [Result] Packer L, Weber SU, Rimbach G. Molecular aspects of alpha-tocotrienol antioxidant action and cell signalling. J Nutr. 2001 Feb;131(2):369S-73S. doi: 10.1093/jn/131.2.369S. PMID 11160563
- [Result] Houston MC, Fazio S, Chilton FH, Wise DE, Jones KB, Barringer TA, Bramlet DA. Nonpharmacologic treatment of dyslipidemia. Prog Cardiovasc Dis. 2009 Sep-Oct;52(2):61-94. doi: 10.1016/j.pcad.2009.02.002. No abstract available. PMID 19732602
- [Result] Zaiden N, Yap WN, Ong S, Xu CH, Teo VH, Chang CP, Zhang XW, Nesaretnam K, Shiba S, Yap YL. Gamma delta tocotrienols reduce hepatic triglyceride synthesis and VLDL secretion. J Atheroscler Thromb. 2010 Oct 27;17(10):1019-32. doi: 10.5551/jat.4911. Epub 2010 Aug 10. PMID 20702976
- [Result] Qureshi AA, Sami SA, Salser WA, Khan FA. Synergistic effect of tocotrienol-rich fraction (TRF(25)) of rice bran and lovastatin on lipid parameters in hypercholesterolemic humans. J Nutr Biochem. 2001 Jun;12(6):318-329. doi: 10.1016/s0955-2863(01)00144-9. PMID 11516635
- [Result] Qureshi AA, Sami SA, Salser WA, Khan FA. Dose-dependent suppression of serum cholesterol by tocotrienol-rich fraction (TRF25) of rice bran in hypercholesterolemic humans. Atherosclerosis. 2002 Mar;161(1):199-207. doi: 10.1016/s0021-9150(01)00619-0. PMID 11882333
- [Result] Qureshi AA, Sami SA, Khan FA. Effects of stabilized rice bran, its soluble and fiber fractions on blood glucose levels and serum lipid parameters in humans with diabetes mellitus Types I and II. J Nutr Biochem. 2002 Mar;13(3):175-187. doi: 10.1016/s0955-2863(01)00211-x. PMID 11893482
- [Result] Montonen J, Knekt P, Jarvinen R, Reunanen A. Dietary antioxidant intake and risk of type 2 diabetes. Diabetes Care. 2004 Feb;27(2):362-6. doi: 10.2337/diacare.27.2.362. PMID 14747214
- [Result] Baliarsingh S, Beg ZH, Ahmad J. The therapeutic impacts of tocotrienols in type 2 diabetic patients with hyperlipidemia. Atherosclerosis. 2005 Oct;182(2):367-74. doi: 10.1016/j.atherosclerosis.2005.02.020. Epub 2005 Apr 20. PMID 16159610
- [Result] Ford ES. Prevalence of the metabolic syndrome defined by the International Diabetes Federation among adults in the U.S. Diabetes Care. 2005 Nov;28(11):2745-9. doi: 10.2337/diacare.28.11.2745. PMID 16249550
- [Result] Wilson PW, D'Agostino RB, Parise H, Sullivan L, Meigs JB. Metabolic syndrome as a precursor of cardiovascular disease and type 2 diabetes mellitus. Circulation. 2005 Nov 15;112(20):3066-72. doi: 10.1161/CIRCULATIONAHA.105.539528. Epub 2005 Nov 7. PMID 16275870
- [Result] Miyazawa T, Shibata A, Sookwong P, Kawakami Y, Eitsuka T, Asai A, Oikawa S, Nakagawa K. Antiangiogenic and anticancer potential of unsaturated vitamin E (tocotrienol). J Nutr Biochem. 2009 Feb;20(2):79-86. doi: 10.1016/j.jnutbio.2008.09.003. Epub 2008 Dec 13. PMID 19071006
- [Result] Shibata A, Nakagawa K, Sookwong P, Tsuzuki T, Oikawa S, Miyazawa T. Tumor anti-angiogenic effect and mechanism of action of delta-tocotrienol. Biochem Pharmacol. 2008 Aug 1;76(3):330-9. doi: 10.1016/j.bcp.2008.05.017. Epub 2008 May 28. PMID 18599020
- [Result] Shibata A, Nakagawa K, Sookwong P, Tsuduki T, Oikawa S, Miyazawa T. delta-Tocotrienol suppresses VEGF induced angiogenesis whereas alpha-tocopherol does not. J Agric Food Chem. 2009 Sep 23;57(18):8696-704. doi: 10.1021/jf9012899. PMID 19702331
- [Result] Qureshi AA, Qureshi N, Hasler-Rapacz JO, Weber FE, Chaudhary V, Crenshaw TD, Gapor A, Ong AS, Chong YH, Peterson D. Dietary tocotrienols reduce concentrations of plasma cholesterol, apolipoprotein B, thromboxane B2, and platelet factor 4 in pigs with inherited hyperlipidemias. Am J Clin Nutr. 1991 Apr;53(4 Suppl):1042S-1046S. doi: 10.1093/ajcn/53.4.1042S. PMID 2012015
- [Result] Naito Y, Shimozawa M, Kuroda M, Nakabe N, Manabe H, Katada K, Kokura S, Ichikawa H, Yoshida N, Noguchi N, Yoshikawa T. Tocotrienols reduce 25-hydroxycholesterol-induced monocyte-endothelial cell interaction by inhibiting the surface expression of adhesion molecules. Atherosclerosis. 2005 May;180(1):19-25. doi: 10.1016/j.atherosclerosis.2004.11.017. Epub 2005 Jan 12. PMID 15823271
- [Result] Campbell LA, Kuo CC. Chlamydia pneumoniae--an infectious risk factor for atherosclerosis? Nat Rev Microbiol. 2004 Jan;2(1):23-32. doi: 10.1038/nrmicro796. PMID 15035006
- [Result] Yamada Y, Obayashi M, Ishikawa T, Kiso Y, Ono Y, Yamashita K. Dietary tocotrienol reduces UVB-induced skin damage and sesamin enhances tocotrienol effects in hairless mice. J Nutr Sci Vitaminol (Tokyo). 2008 Apr;54(2):117-23. doi: 10.3177/jnsv.54.117. PMID 18490840
- [Result] Michihara A, Ogawa S, Kamizaki Y, Akasaki K. Effect of delta-tocotrienol on melanin content and enzymes for melanin synthesis in mouse melanoma cells. Biol Pharm Bull. 2010;33(9):1471-6. doi: 10.1248/bpb.33.1471. PMID 20823559
- [Result] Traber MG, Podda M, Weber C, Thiele J, Rallis M, Packer L. Diet-derived and topically applied tocotrienols accumulate in skin and protect the tissue against ultraviolet light-induced oxidative stress. Asia Pac J Clin Nutr. 1997 Mar;6(1):63-7. PMID 24394657
- [Result] Sen CK, Khanna S, Roy S. Tocotrienols: Vitamin E beyond tocopherols. Life Sci. 2006 Mar 27;78(18):2088-98. doi: 10.1016/j.lfs.2005.12.001. Epub 2006 Feb 3. PMID 16458936
- [Result] Husain K, Francois RA, Hutchinson SZ, Neuger AM, Lush R, Coppola D, Sebti S, Malafa MP. Vitamin E delta-tocotrienol levels in tumor and pancreatic tissue of mice after oral administration. Pharmacology. 2009;83(3):157-63. doi: 10.1159/000190792. Epub 2009 Jan 13. PMID 19142032
- [Result] Hussein D, Mo H. d-delta-Tocotrienol-mediated suppression of the proliferation of human PANC-1, MIA PaCa-2, and BxPC-3 pancreatic carcinoma cells. Pancreas. 2009 May;38(4):e124-36. doi: 10.1097/MPA.0b013e3181a20f9c. PMID 19346993
- [Result] Husain K, Francois RA, Yamauchi T, Perez M, Sebti SM, Malafa MP. Vitamin E delta-tocotrienol augments the antitumor activity of gemcitabine and suppresses constitutive NF-kappaB activation in pancreatic cancer. Mol Cancer Ther. 2011 Dec;10(12):2363-72. doi: 10.1158/1535-7163.MCT-11-0424. Epub 2011 Oct 4. PMID 21971120
- [Result] Palapattu GS, Sutcliffe S, Bastian PJ, Platz EA, De Marzo AM, Isaacs WB, Nelson WG. Prostate carcinogenesis and inflammation: emerging insights. Carcinogenesis. 2005 Jul;26(7):1170-81. doi: 10.1093/carcin/bgh317. Epub 2004 Oct 21. PMID 15498784
- [Result] Lippman SM, Klein EA, Goodman PJ, Lucia MS, Thompson IM, Ford LG, Parnes HL, Minasian LM, Gaziano JM, Hartline JA, Parsons JK, Bearden JD 3rd, Crawford ED, Goodman GE, Claudio J, Winquist E, Cook ED, Karp DD, Walther P, Lieber MM, Kristal AR, Darke AK, Arnold KB, Ganz PA, Santella RM, Albanes D, Taylor PR, Probstfield JL, Jagpal TJ, Crowley JJ, Meyskens FL Jr, Baker LH, Coltman CA Jr. Effect of selenium and vitamin E on risk of prostate cancer and other cancers: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2009 Jan 7;301(1):39-51. doi: 10.1001/jama.2008.864. Epub 2008 Dec 9. PMID 19066370
- [Result] Klein EA, Thompson IM Jr, Tangen CM, Crowley JJ, Lucia MS, Goodman PJ, Minasian LM, Ford LG, Parnes HL, Gaziano JM, Karp DD, Lieber MM, Walther PJ, Klotz L, Parsons JK, Chin JL, Darke AK, Lippman SM, Goodman GE, Meyskens FL Jr, Baker LH. Vitamin E and the risk of prostate cancer: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2011 Oct 12;306(14):1549-56. doi: 10.1001/jama.2011.1437. PMID 21990298
- [Result] Ji X, Wang Z, Geamanu A, Sarkar FH, Gupta SV. Inhibition of cell growth and induction of apoptosis in non-small cell lung cancer cells by delta-tocotrienol is associated with notch-1 down-regulation. J Cell Biochem. 2011 Oct;112(10):2773-83. doi: 10.1002/jcb.23184. PMID 21598300
- [Result] Yano Y, Satoh H, Fukumoto K, Kumadaki I, Ichikawa T, Yamada K, Hagiwara K, Yano T. Induction of cytotoxicity in human lung adenocarcinoma cells by 6-O-carboxypropyl-alpha-tocotrienol, a redox-silent derivative of alpha-tocotrienol. Int J Cancer. 2005 Jul 10;115(5):839-46. doi: 10.1002/ijc.20809. PMID 15723336
- [Result] Zhang JS, Li DM, He N, Liu YH, Wang CH, Jiang SQ, Chen BQ, Liu JR. A paraptosis-like cell death induced by delta-tocotrienol in human colon carcinoma SW620 cells is associated with the suppression of the Wnt signaling pathway. Toxicology. 2011 Jul 11;285(1-2):8-17. doi: 10.1016/j.tox.2011.03.011. Epub 2011 Mar 29. PMID 21453743
- [Result] Xu WL, Liu JR, Liu HK, Qi GY, Sun XR, Sun WG, Chen BQ. Inhibition of proliferation and induction of apoptosis by gamma-tocotrienol in human colon carcinoma HT-29 cells. Nutrition. 2009 May;25(5):555-66. doi: 10.1016/j.nut.2008.10.019. Epub 2009 Jan 3. PMID 19121919
- [Result] Gillen CD, Walmsley RS, Prior P, Andrews HA, Allan RN. Ulcerative colitis and Crohn's disease: a comparison of the colorectal cancer risk in extensive colitis. Gut. 1994 Nov;35(11):1590-2. doi: 10.1136/gut.35.11.1590. PMID 7828978
- [Result] Shibata A, Nakagawa K, Sookwong P, Tsuduki T, Asai A, Miyazawa T. alpha-Tocopherol attenuates the cytotoxic effect of delta-tocotrienol in human colorectal adenocarcinoma cells. Biochem Biophys Res Commun. 2010 Jun 25;397(2):214-9. doi: 10.1016/j.bbrc.2010.05.087. Epub 2010 May 20. PMID 20493172
- [Result] Sun W, Wang Q, Chen B, Liu J, Liu H, Xu W. Gamma-tocotrienol-induced apoptosis in human gastric cancer SGC-7901 cells is associated with a suppression in mitogen-activated protein kinase signalling. Br J Nutr. 2008 Jun;99(6):1247-54. doi: 10.1017/S0007114507879128. Epub 2007 Dec 17. PMID 18081943
- [Result] Nesaretnam K, Stephen R, Dils R, Darbre P. Tocotrienols inhibit the growth of human breast cancer cells irrespective of estrogen receptor status. Lipids. 1998 May;33(5):461-9. doi: 10.1007/s11745-998-0229-3. PMID 9625593
- [Result] Nesaretnam K, Meganathan P, Veerasenan SD, Selvaduray KR. Tocotrienols and breast cancer: the evidence to date. Genes Nutr. 2012 Jan;7(1):3-9. doi: 10.1007/s12263-011-0224-z. Epub 2011 Apr 24. PMID 21516480
- [Result] Shun MC, Yu W, Gapor A, Parsons R, Atkinson J, Sanders BG, Kline K. Pro-apoptotic mechanisms of action of a novel vitamin E analog (alpha-TEA) and a naturally occurring form of vitamin E (delta-tocotrienol) in MDA-MB-435 human breast cancer cells. Nutr Cancer. 2004;48(1):95-105. doi: 10.1207/s15327914nc4801_13. PMID 15203383
- [Result] Guthrie N, Gapor A, Chambers AF, Carroll KK. Inhibition of proliferation of estrogen receptor-negative MDA-MB-435 and -positive MCF-7 human breast cancer cells by palm oil tocotrienols and tamoxifen, alone and in combination. J Nutr. 1997 Mar;127(3):544S-548S. doi: 10.1093/jn/127.3.544S. PMID 9082043
- [Result] McIntyre BS, Briski KP, Gapor A, Sylvester PW. Antiproliferative and apoptotic effects of tocopherols and tocotrienols on preneoplastic and neoplastic mouse mammary epithelial cells. Proc Soc Exp Biol Med. 2000 Sep;224(4):292-301. doi: 10.1046/j.1525-1373.2000.22434.x. PMID 10964265
- [Result] Sylvester PW, Shah SJ. Mechanisms mediating the antiproliferative and apoptotic effects of vitamin E in mammary cancer cells. Front Biosci. 2005 Jan 1;10:699-709. doi: 10.2741/1565. Print 2005 Jan 1. PMID 15569611
- [Result] Shah S, Gapor A, Sylvester PW. Role of caspase-8 activation in mediating vitamin E-induced apoptosis in murine mammary cancer cells. Nutr Cancer. 2003;45(2):236-46. doi: 10.1207/S15327914NC4502_14. PMID 12881019
- [Result] Takahashi K, Loo G. Disruption of mitochondria during tocotrienol-induced apoptosis in MDA-MB-231 human breast cancer cells. Biochem Pharmacol. 2004 Jan 15;67(2):315-24. doi: 10.1016/j.bcp.2003.07.015. PMID 14698044
- [Result] Nesaretnam K, Ambra R, Selvaduray KR, Radhakrishnan A, Canali R, Virgili F. Tocotrienol-rich fraction from palm oil and gene expression in human breast cancer cells. Ann N Y Acad Sci. 2004 Dec;1031:143-57. doi: 10.1196/annals.1331.014. PMID 15753141
- [Result] Shah SJ, Sylvester PW. Gamma-tocotrienol inhibits neoplastic mammary epithelial cell proliferation by decreasing Akt and nuclear factor kappaB activity. Exp Biol Med (Maywood). 2005 Apr;230(4):235-41. doi: 10.1177/153537020523000402. PMID 15792944
- [Result] Shah SJ, Sylvester PW. Tocotrienol-induced cytotoxicity is unrelated to mitochondrial stress apoptotic signaling in neoplastic mammary epithelial cells. Biochem Cell Biol. 2005 Feb;83(1):86-95. doi: 10.1139/o04-127. PMID 15746970
- [Result] Samant GV, Sylvester PW. gamma-Tocotrienol inhibits ErbB3-dependent PI3K/Akt mitogenic signalling in neoplastic mammary epithelial cells. Cell Prolif. 2006 Dec;39(6):563-74. doi: 10.1111/j.1365-2184.2006.00412.x. PMID 17109639
- [Result] Sylvester PW, Shah SJ, Samant GV. Intracellular signaling mechanisms mediating the antiproliferative and apoptotic effects of gamma-tocotrienol in neoplastic mammary epithelial cells. J Plant Physiol. 2005 Jul;162(7):803-10. doi: 10.1016/j.jplph.2005.04.014. PMID 16008108
- [Result] Weber C, Podda M, Rallis M, Thiele JJ, Traber MG, Packer L. Efficacy of topically applied tocopherols and tocotrienols in protection of murine skin from oxidative damage induced by UV-irradiation. Free Radic Biol Med. 1997;22(5):761-9. doi: 10.1016/s0891-5849(96)00346-2. PMID 9119243
- [Result] He L, Mo H, Hadisusilo S, Qureshi AA, Elson CE. Isoprenoids suppress the growth of murine B16 melanomas in vitro and in vivo. J Nutr. 1997 May;127(5):668-74. doi: 10.1093/jn/127.5.668. PMID 9164984
- [Result] Mensink RP, van Houwelingen AC, Kromhout D, Hornstra G. A vitamin E concentrate rich in tocotrienols had no effect on serum lipids, lipoproteins, or platelet function in men with mildly elevated serum lipid concentrations. Am J Clin Nutr. 1999 Feb;69(2):213-9. doi: 10.1093/ajcn/69.2.213. PMID 9989682
- [Result] Newaz MA, Nawal NN. Effect of gamma-tocotrienol on blood pressure, lipid peroxidation and total antioxidant status in spontaneously hypertensive rats (SHR). Clin Exp Hypertens. 1999 Nov;21(8):1297-313. doi: 10.3109/10641969909070850. PMID 10574414
- [Result] Newaz MA, Yousefipour Z, Nawal N, Adeeb N. Nitric oxide synthase activity in blood vessels of spontaneously hypertensive rats: antioxidant protection by gamma-tocotrienol. J Physiol Pharmacol. 2003 Sep;54(3):319-27. PMID 14566071
- [Result] Pearson CK, Barnes MM. The absorption and distribution of the naturally occurring tocochromanols in he rat. Br J Nutr. 1970 Jun;24(2):581-7. doi: 10.1079/bjn19700056. No abstract available. PMID 5452708
- [Result] Yap SP, Yuen KH, Wong JW. Pharmacokinetics and bioavailability of alpha-, gamma- and delta-tocotrienols under different food status. J Pharm Pharmacol. 2001 Jan;53(1):67-71. doi: 10.1211/0022357011775208. PMID 11206194
- [Result] Yu W, Simmons-Menchaca M, Gapor A, Sanders BG, Kline K. Induction of apoptosis in human breast cancer cells by tocopherols and tocotrienols. Nutr Cancer. 1999;33(1):26-32. doi: 10.1080/01635589909514744. PMID 10227040
- [Result] Elangovan S, Hsieh TC, Wu JM. Growth inhibition of human MDA-mB-231 breast cancer cells by delta-tocotrienol is associated with loss of cyclin D1/CDK4 expression and accompanying changes in the state of phosphorylation of the retinoblastoma tumor suppressor gene product. Anticancer Res. 2008 Sep-Oct;28(5A):2641-7. PMID 19035289
- [Result] Pierpaoli E, Viola V, Pilolli F, Piroddi M, Galli F, Provinciali M. Gamma- and delta-tocotrienols exert a more potent anticancer effect than alpha-tocopheryl succinate on breast cancer cell lines irrespective of HER-2/neu expression. Life Sci. 2010 Apr 24;86(17-18):668-75. doi: 10.1016/j.lfs.2010.02.018. Epub 2010 Feb 25. PMID 20188744
- [Result] Viola V, Ciffolilli S, Legnaioli S, Piroddi M, Betti M, Mazzini F, Pierpaoli E, Provinciali M, Galli F. Mitochondrial-dependent anticancer activity of delta-tocotrienol and its synthetic derivatives in HER-2/neu overexpressing breast adenocarcinoma cells. Biofactors. 2013 Jul-Aug;39(4):485-93. doi: 10.1002/biof.1089. Epub 2013 Jan 30. PMID 23361894
- [Result] Comitato R, Leoni G, Canali R, Ambra R, Nesaretnam K, Virgili F. Tocotrienols activity in MCF-7 breast cancer cells: involvement of ERbeta signal transduction. Mol Nutr Food Res. 2010 May;54(5):669-78. doi: 10.1002/mnfr.200900383. PMID 20306477
- [Result] Comitato R, Nesaretnam K, Leoni G, Ambra R, Canali R, Bolli A, Marino M, Virgili F. A novel mechanism of natural vitamin E tocotrienol activity: involvement of ERbeta signal transduction. Am J Physiol Endocrinol Metab. 2009 Aug;297(2):E427-37. doi: 10.1152/ajpendo.00187.2009. Epub 2009 Jun 2. PMID 19491296
- [Result] Sylvester PW, Akl MR, Malaviya A, Parajuli P, Ananthula S, Tiwari RV, Ayoub NM. Potential role of tocotrienols in the treatment and prevention of breast cancer. Biofactors. 2014 Jan-Feb;40(1):49-58. doi: 10.1002/biof.1116. Epub 2013 Jun 27. PMID 23804535
- [Result] Nesaretnam K, Selvaduray KR, Abdul Razak G, Veerasenan SD, Gomez PA. Effectiveness of tocotrienol-rich fraction combined with tamoxifen in the management of women with early breast cancer: a pilot clinical trial. Breast Cancer Res. 2010;12(5):R81. doi: 10.1186/bcr2726. Epub 2010 Oct 8. PMID 20929592
- [Result] Howe GR, Hirohata T, Hislop TG, Iscovich JM, Yuan JM, Katsouyanni K, Lubin F, Marubini E, Modan B, Rohan T, et al. Dietary factors and risk of breast cancer: combined analysis of 12 case-control studies. J Natl Cancer Inst. 1990 Apr 4;82(7):561-9. doi: 10.1093/jnci/82.7.561. PMID 2156081
- [Result] Sestak I, Distler W, Forbes JF, Dowsett M, Howell A, Cuzick J. Effect of body mass index on recurrences in tamoxifen and anastrozole treated women: an exploratory analysis from the ATAC trial. J Clin Oncol. 2010 Jul 20;28(21):3411-5. doi: 10.1200/JCO.2009.27.2021. Epub 2010 Jun 14. PMID 20547990
- [Result] Sieri S, Pala V, Brighenti F, Agnoli C, Grioni S, Berrino F, Scazzina F, Palli D, Masala G, Vineis P, Sacerdote C, Tumino R, Giurdanella MC, Mattiello A, Panico S, Krogh V. High glycemic diet and breast cancer occurrence in the Italian EPIC cohort. Nutr Metab Cardiovasc Dis. 2013 Jul;23(7):628-34. doi: 10.1016/j.numecd.2012.01.001. Epub 2012 Apr 10. PMID 22497978
- [Result] Pasanisi P, Berrino F, De Petris M, Venturelli E, Mastroianni A, Panico S. Metabolic syndrome as a prognostic factor for breast cancer recurrences. Int J Cancer. 2006 Jul 1;119(1):236-8. doi: 10.1002/ijc.21812. PMID 16450399
- [Result] Villarini A, Pasanisi P, Traina A, Mano MP, Bonanni B, Panico S, Scipioni C, Galasso R, Paduos A, Simeoni M, Bellotti E, Barbero M, Macellari G, Venturelli E, Raimondi M, Bruno E, Gargano G, Fornaciari G, Morelli D, Seregni E, Krogh V, Berrino F. Lifestyle and breast cancer recurrences: the DIANA-5 trial. Tumori. 2012 Jan-Feb;98(1):1-18. doi: 10.1177/030089161209800101. PMID 22495696
- [Result] Wiseman M. The second World Cancer Research Fund/American Institute for Cancer Research expert report. Food, nutrition, physical activity, and the prevention of cancer: a global perspective. Proc Nutr Soc. 2008 Aug;67(3):253-6. doi: 10.1017/S002966510800712X. Epub 2008 May 1. PMID 18452640
- [Result] Donini LM, Cuzzolaro M, Spera G, Badiali M, Basso N, Bollea MR, Bosello O, Brunani A, Busetto L, Cairella G, Cannella C, Capodaglio P, Carbonelli MG, Castellaneta E, Castra R, Clini E, Contaldo F, Dalla Ragione L, Dalle Grave R, D'Andrea F, Del Balzo V, De Cristofaro P, Di Flaviano E, Fassino S, Ferro AM, Forestieri P, Franzoni E, Gentile MG, Giustini A, Jacoangeli F, Lubrano C, Lucchin L, Manara F, Marangi G, Marcelli M, Marchesini G, Marri G, Marrocco W, Melchionda N, Mezzani B, Migliaccio P, Muratori F, Nizzoli U, Ostuzzi R, Panzolato G, Pasanisi F, Persichetti P, Petroni ML, Pontieri V, Prosperi E, Renna C, Rovera G, Santini F, Saraceni V, Savina C, Scuderi N, Silecchia G, Strollo F, Todisco P, Tubili C, Ugolini G, Zamboni M. [Obesity and Eating Disorders. Indications for the different levels of care. An Italian Expert Consensus Document]. Eat Weight Disord. 2010 Mar-Jun;15(1-2 Suppl):1-31. Italian. PMID 20975326